The Effect of Guided İmagery Applied Before and After Surgery on Surgical Anxiety, Pain and Analgesic Consumption in Patients Undergoing Total Joint Arthroplasty: A Randomized Controlled Trial Study Protocol and Statistical Analysis of a Randomized Controlled Trial

## The Effect of Guided İmagery Applied Before and After Surgery on Surgical Anxiety, Pain and Analgesic Consumption in Patients Undergoing Total Joint Arthroplasty: A Randomized Controlled Trial Study Protocol and Statistical Analysis of a Randomized Controlled Trial



The statistical analyses of the study will be performed using the SPSS 29.0 and R-Studio software packages. Descriptive statistics for the qualitative variables included in the study will be presented as frequencies and percentages, while quantitative variables will be presented as means, standard deviations, medians, minimum, and maximum values. The normality of quantitative variables will be examined using the Shapiro Wilk test. Independent sample t-tests and Mann Whitney U tests will be used for independent group comparisons of variables, while dependent sample t-tests and Wilcoxon tests will be used for dependent group comparisons. Relationships between quantitative variables will be evaluated using Pearson and Spearman correlation coefficients. Relationships between quantitative variables will be evaluated using Pearson and Spearman correlation coefficients. In all statistical comparisons in the study, results with a p-value below 0.05 will be considered statistically significant.